CLINICAL TRIAL: NCT04649242
Title: Phase 3, Multicenter, Randomized, Double-blind, Group Sequential, Placebo-controlled Study to Assess Efficacy and Safety of Rimegepant for the Treatment of Migraine (With or Without Aura) in Children and Adolescents ≥ 6 to < 18 Years of Age
Brief Title: Randomized Study in Children and Adolescents With Migraine: Acute Treatment
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BHV3000-311; C4951002 (Other: Alias Study Number); 2020-003517-35 (Registry Identifier: CTIS (EU)); 2024-512743-23-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2020-11-23; First posted 2020-12-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Migraine
Keywords: Migraine; Acute treatment; Phonophobia; Photophobia; Nausea; Pediatric; Children; Adolescent; Pediatric Migraine
MeSH Terms: conditions — Migraine Disorders; Hyperacusis; Photophobia; Nausea | interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV3000 (active drug) (Active Comparator): BHV3000 (rimegepant) 75 mg or 50 mg ODT
  Interventions: Drug: Rimegepant/BHV3000
- Placebo (Placebo Comparator): Matching 75 mg or 50 mg ODT placebo
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: Rimegepant/BHV3000 — BHV3000 (rimegepant) 75 mg or 50 mg ODT
  Arms: BHV3000 (active drug)
Drug: Matching placebo — Matching 75 mg or 50 mg ODT placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the safety and efficacy of BHV-3000 versus placebo in the acute treatment of moderate or severe migraine in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. History of migraine (with or without aura) for > 6 months before Screening according to the IHS Classification ICHD-319 specifications for pediatric migraine. History may be verified using both medical records and recall by the participant and/or participant's parent(s)/legal representative(s).
2. History of 1 to 8 moderate or severe attacks per month during the 2 months prior to enrollment, with attacks lasting > 3 hours without treatment, and attacks occurring at intervals > 24 hours.
3. Prophylactic migraine medication are permitted if the dose has been stable for at least 12 weeks prior to the Baseline Visit, and the dose is not expected to change during the course of the study.

   1. Participants may remain on one (1) medication with possible migraine prophylactic effects, excluding CGRP antagonists [biologic or small molecule], during the treatment phases.
   2. Concomitant use of a CGRP antagonist, such as erenumab or fremanezumab, is prohibited.
   3. Previously discontinued prophylactic migraine medication must have done so at least 90 days prior to the Screening Visit.
4. Verbally distinguish between migraine and other types of headaches.
5. Participants must have a weight > 40 kg at the Screening Visit.
6. Adequate venous access for blood sampling.
7. Male and female participants ≥ 6 to < 18 years of age (participants must not reach their 18th birthday during the study).

Exclusion Criteria:

1. History of cluster headache or hemiplegic migraine headache.
2. Confounding and clinically significant pain syndrome that may interfere with the participant's ability to participate in this study.
3. Current psychiatric condition that is uncontrolled and/or untreated for a minimum of 6 months prior to the Screening Visit. Participants with a lifetime history of psychosis and/or mania.
4. History of suicidal behavior or major psychiatric disorder.
5. Current diagnosis or history of substance abuse; positive drug test at Screening.
6. History of moderate or severe head trauma or other neurological disorder (including seizure disorder) or systemic medical disease that is likely to affect central nervous system functioning.
7. Recent or planned surgery, requiring general anesthesia, <8 weeks prior to the Screening Visit.
8. Participant has had gastrointestinal surgery that interferes with physiological absorption and motility (i.e., gastric bypass, duodenectomy, or gastric banding).
9. Current diagnosis of viral hepatitis or a history of liver disease.
10. Conditions considered clinically relevant in the context of the study such as uncontrolled hypertension (high blood pressure), diabetes, a life-threatening allergy

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2100 (Estimated)
Dates: Start 2021-01-15 (Actual); Primary Completion 2029-01-09 (Estimated); Study Completion 2029-01-09 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of rimegepant compared with placebo in the acute treatment of migraine in adolescent population (≥ 12 to <18 years of age) as measured by pain freedom using the number of patients reporting no pain. | 2 hours post-dose
  Pain freedom will be assessed in adolescent population (≥ 12 to < 18 years of age) on a 4-point numeric rating scale (0=none, 1=mild, 2=moderate, 3=severe).

SECONDARY OUTCOMES:
To compare rimegepant with placebo for pain freedom in children and adolescents combined. | 2 hours post-dose
  Pain freedom will be assessed in children and adolescents (≥ 6 to < 18 years of age) using a 4-point numeric rating scale (0=none, 1=mild, 2=moderate, 3=severe).
  Pain freedom will be assessed in children (> 6 to < 12 years of age) using the 5-Face VAS (Face 5 = 'severe pain', Faces 4 and 3 = 'moderate pain', Face 2 = 'mild pain', Face 1 = 'no pain').
To compare rimegepant with placebo on freedom from the most bothersome symptom (MBS) associated with migraine in adolescents. | 2 hours post-dose
  Freedom from MBS (nausea, phonophobia or photophobia) will be measured using a binary scale (0=absent, 1=present).
To compare rimegepant with placebo on the probabilities of requiring rescue medication within in adolescents. | Within 24 hours and 48 hours of initial treatment
  Use of rescue medication will be assessed using the numbers of participants that take rescue medication.
To compare rimegepant with placebo on sustained pain freedom in adolescents. | 2 to 24 hours post-dose
  Sustained pain freedom will be assessed using the number of participants that do not use any rescue medications and do not experience any headache pain post dose.
To compare rimegepant with placebo on sustained pain freedom in adolescents. | 2 to 48 hours post-dose
  Sustained pain freedom will be assessed using the number of participants that do not use any rescue medications and do not experience any headache pain post dose.
To compare rimegepant with placebo on the ability to function normally as reported on the Functional Disability scale in adolescents. | 2 hours post-dose
  The proportion of participants able to function normally will be assessed using the number that self-report as "normal" on the Functional Disability scale.
To compare rimegepant with placebo for pain freedom in children. | 2 hours post-dose
  Pain freedom will be assessed using the number of children (≥ 6 to < 12 years of age) that report no pain measured by a 5-Face VAS (Face 5 = 'severe pain', Faces 4 and 3 = 'moderate pain', Face 2 = 'mild pain', Face 1 = 'no pain').
To compare rimegepant with placebo on freedom from the most bothersome symptom (MBS) associated with migraine in children and combined children and adolescents. | 2 hours post-dose
  Freedom from the most bothersome symptom (nausea, phonophobia or photophobia) will be assessed using the number of participants that report the absence of MBS measured using a binary scale (0=absent, 1=present).
To compare rimegepant with placebo on the probabilities of requiring rescue medication in children and combined children and adolescents. | Within 24 hours and 48 hours of initial treatment.
  The probabilities of requiring rescue medication will be assessed using the numbers of participants that take rescue medication within initial treatment.
To compare rimegepant with placebo on sustained pain freedom in children and combined children and adolescents. | 2 to 24 hours post-dose
  Sustained pain freedom will be assessed using the number of participants that do not use any rescue medications and do not experience any headache pain post dose.
To compare rimegepant with placebo on sustained pain freedom in children and combined children and adolescents. | 2 to 48 hours post-dose
  Sustained pain freedom will be assessed using the number of participants that do not use any rescue medications and do not experience any headache pain post dose.
To compare rimegepant with placebo on freedom from photophobia in adolescents, children and combined children and adolescents. | 2 hours post-dose
  Freedom from photophobia will be assessed by the number of participants that report the absence of photophobia post dose that reported the presence of photophobia at baseline.
To compare rimegepant with placebo on freedom from phonophobia in adolescents, children and combined children and adolescents. | 2 hours post-dose
  Freedom from phonophobia will be assessed by the number of participants that report the absence of phonophobia post dose that reported the presence of phonophobia at baseline.
To compare rimegepant with placebo on freedom from nausea in adolescents, children and combined children and adolescents. | 2 hours post-dose
  Freedom from nausea will be assessed by the number of participants that report the absence of nausea post dose that reported the presence of nausea at baseline.
To compare rimegepant with placebo on pain relief in adolescents, children and combined children and adolescents. | 2 hours post-dose
  Pain relief will be assessed using the number of participants that report a pain level of moderate or severe at baseline and then report a pain level of none or mild post dose.
To compare rimegepant with placebo in adolescents, children and combined children and adolescents on pain relief. | Time to patients first report of pain relief of none or mild post dose up to 48 hours.
  Time to first report of pain relief will be based on the first time point a participant reports a pain level of none or mild.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (242):
- United States (166):
  - Achieve Clinical Research, LLC d/b/a Accel Research Sites-Neurology and Neurodiagnostic of Alabama, Birmingham, Alabama
  - Perseverance Research Center, LLC, Scottsdale, Arizona
  - Physicians Research Group, Tempe, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - Adult & Child Neurology Medical Associates, Costa Mesa, California
  - ProScience Research Group, Culver City, California
  - Memorial Health Services, Fountain Valley, California
  - Neuro-Pain Medical Center, Fresno, California
  - Altman Clinical and Translational Research Institute-IDS, La Jolla, California
  - University of California, San Diego Altman Clinical Translational Research Institute, La Jolla, California
  - Adult & Child Neurology Medical Associates, Long Beach, California
  - Miller Children's & Women's Hospital Long Beach, Long Beach, California
  - National Research Institute, Los Angeles, California
  - Velocity Clinical Research - North Hollywood, North Hollywood, California
  - Children's Hospital of Orange County - Inpatient Pharmacy, Orange, California
  - Children's Hospital of Orange County - Neuroscience Center, Orange, California
  - Children's Hospital of Orange County, Orange, California
  - The Neurology Group, Pomona, California
  - University of California, Davis Midtown Clinic, Sacramento, California
  - UC Davis Medical Center, Investigational Drug Service (IDS) Pharmacy, Sacramento, California
  - University of California, Davis Clinical and Translational Science Center Clinical Research (CCRC), Sacramento, California
  - Velocity Clinical Research, San Bernardino (IP Delivery and Administering Location), San Bernardino, California
  - Pacific Clinical Research Management Group LLC, Upland, California
  - Sunwise Clinical Research, Walnut Creek, California
  - Children's Hospital Colorado- lnvestigational Drug Services, Aurora, Colorado
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado Springs Neurological Associates, PC, Colorado Springs, Colorado
  - CT Clinical Research, Cromwell, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Ki Health Partners, LLc, dba New England Institute for Clinical Research, Stamford, Connecticut
  - Nemours Children's Hospital, Delaware, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Topaz Clinical Research, Inc., Apopka, Florida
  - Beautiful Minds Clinical Research Center, Cutler Bay, Florida
  - DeLand Clinical Research Unit, DeLand, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Watson Clinic Center for Research, Inc., Lakeland, Florida
  - Watson Clinic LLP, Lakeland, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - Medical Research Center of Miami II, Inc, Miami, Florida
  - Nicklaus Children's Hospital, Research Institute, Miami, Florida
  - Brainstorm Research, Miami, Florida
  - South Florida Research Phase I-IV, Inc, Miami Springs, Florida
  - Advanced Research for Health Improvement, LLC/ Dr. Cordero's Pediatric Office, Naples, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Coastal Clinical Research Specialists, Orange Park, Florida
  - Clinical Associates of Orlando, LLC, Orlando, Florida
  - Bioresearch Institute, Pembroke Pines, Florida
  - Forcare Clinical Research, Tampa, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Children's Healthcare of Atlanta, Inc., Atlanta, Georgia
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Pivotal Clinical Research & Associates, LLC, Brunswick, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Chicago Headache Center & Research Institute, Chicago, Illinois
  - AMR-Baber Research Inc, Naperville, Illinois
  - Options Research Group, LLC, Westfield, Indiana
  - Meridian Clinical Research, LLC, Sioux City, Iowa
  - Integrated Clinical Trial Services, West Des Moines, Iowa
  - Clinical Associates Midwest, LLC, Kansas City, Kansas
  - College Park Family Care Center Physicians Group- Neurology Research Dept., Overland Park, Kansas
  - Kentucky Neuroscience Institute Child Neurology-- "Patients Seen", Lexington, Kentucky
  - UK Center for Clinical and Translational Science (CCTS) -- "Patients Seen", Lexington, Kentucky
  - University of Kentucky Hospital, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Neurology and Headache Center, Inc., Shreveport, Louisiana
  - Boston Clinical Trials, Boston, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Michigan Head Pain & Neurological Institute, Ann Arbor, Michigan
  - Corewell Health, for and on behalf of Spectrum Health Hospital and Corewell Health Medical Group, Grand Rapids, Michigan
  - Corewell Health, Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Wellnow Urgent Care and Research, Kalamazoo, Michigan
  - Beaumont Hospital Royal Oak Campus, Royal Oak, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Sharlin Health Neuroscience Research Center, Ozark, Missouri
  - Clinvest Research, LLC, Springfield, Missouri
  - Boeson Research, Great Falls, Montana
  - Boeson Research, Kalispell, Montana
  - Heart & Hands Midwifery, Kalispell, Montana
  - Blue Moose Pediatrics, Missoula, Montana
  - Boeson Research Laboratory, Missoula, Montana
  - Boeson Research, Missoula, Montana
  - Alivation Research, LLC., Lincoln, Nebraska
  - Children's Hospital & Medical Center, Omaha, Nebraska
  - HMH Jersey Shore University Medical Center, Neptune City, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - True North Neurology, Commack, New York
  - Northwell Health/ Division of Pediatric Neurology, Lake Success, New York
  - NYU Langone Hospital-Long Island, Clinical Research Center, Mineola, New York
  - NYU Langone Hospital-Long Island, Pediatric Neurology, Mineola, New York
  - New York Neurology Associates, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Mount Sinai Hospital - Pharmacy Department, New York, New York
  - Columbia University Medical Center Research Pharmacy, New York, New York
  - Columbia University Pediatric Neuromuscular Center, New York, New York
  - Irving Center for Clinical and Translational Research, Outpatient Clinical Research Unit, New York, New York
  - The Neurological Institute of New York, New York, New York
  - The Trustees of Columbia University and The New York and Presbyterian Hospital, New York, New York
  - North Suffolk Neurology P.C, Port Jefferson Station, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Prime Global Research, LLC, The Bronx, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Velocity Clinical Research, Inc., Durham, North Carolina
  - Headache Wellness Center, PC, Greensboro, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Wellnow Urgent Care and Research, Columbus, Ohio
  - Neuro-Behavioral Clinical Research, Inc., North Canton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Lynn Institute of Tulsa, Tulsa, Oklahoma
  - Velocity Clinical Research, Grants Pass, Grants Pass, Oregon
  - Providence Brain & Spine Institute-research coordinator's office, Portland, Oregon
  - Providence Health & Services Investigational Drug Services Westside, Portland, Oregon
  - Providence Pediatric Neurology, Portland, Oregon
  - Clario, Philadelphia, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Velocity Clinical Research-Providence, East Greenwich, Rhode Island
  - Premier Neurology, PC, Greenville, South Carolina
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Velocity Clinical Research - Greenville, Greenville, South Carolina
  - Holston Medical Group., Kingsport, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - Le Bonheur Children's Hospital - Outpatient Building, Memphis, Tennessee
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Le Bonheur Childrens Hospital - Childrens Foundation Research Institute, Memphis, Tennessee
  - Access Clinical Trials, Inc., Nashville, Tennessee
  - Dell Children's Medical Center, Austin, Texas
  - Child Neurology Consultants of Austin - South Austin, Austin, Texas
  - Child Neurology Consultants of Austin - Central Austin, Austin, Texas
  - BioBehavioral Research of Austin, Austin, Texas
  - Houston Clinical Trials, LLC, Bellaire, Texas
  - Infinite Research Group, LLC, Dallas, Texas
  - Children's Medical Center, Dallas, Dallas, Texas
  - Children's Medical Center, Pediatric Anesthesiology Research (Study supplies only), Dallas, Texas
  - Cedar Health Research, Dallas, Texas
  - FutureSearch Trials of Dallas, LLC, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - ANESC Research, El Paso, Texas
  - North Texas Institute of Neurology and Headache, Frisco, Texas
  - UTHealth Houston, Houston, Texas
  - Pain and Headache Centers of Texas, Houston, Texas
  - SCLA Management, Houston, Texas
  - Houston Clinical Research,LLC., Houston, Texas
  - NeuroCare Plus, Houston, Texas
  - AIM Trials, LLC, Plano, Texas
  - JBR Clinical Research, Salt Lake City, Utah
  - Wasatch Clinical Research , LLC(Administrative Location), Salt Lake City, Utah
  - The University of Vermont Medical Center, Burlington, Vermont
  - Pediatric Research of Charlottesville, LLC (Regulatory Only), Charlottesville, Virginia
  - Pediatric Research of Charlottesville, LLC, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Children's Specialty Group, PLLC, Norfolk, Virginia
  - Children's Specialty Group, PLLC, Division of Childhood & Adolescent Neurology, Norfolk, Virginia
  - National Clinical Research, Inc., Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Eastside Therapeutic Resource, Inc. dba Core Clinical Research, Everett, Washington
  - Seattle Children's Hospital Investigational Drug Services, Seattle, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Clinical Investigation Specialists, Inc, Kenosha, Wisconsin
  - University Hospital, Madison, Wisconsin
- Canada (2):
  - OCT Research ULC, Kelowna, British Columbia
  - Diex Recherche Sherbrooke Inc, Sherbrooke, Quebec
- China (38):
  - First Affiliated Hospital of Bengbu Medical College Neurology, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - " The First Affiliated Hospital of Chongqing Medical University", Chongqing, Chongqing Municipality
  - Lanzhou university second hospital, Lanzhou, Gansu
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Jingzhou First People's Hospital, Jingzhou, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Hunan Children's Hospital, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi Children's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Xuzhou Children's Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Hospital of Jilin University, Pediatric Neurology, Changchun, Jilin
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Xi'an Gaoxin Hospital Neurology Department, Xi'an, Shaanxi
  - Yan 'an University Xianyang Hospital, Xianyang, Shaanxi
  - Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ningbo Women and Children's Hospital, Ningbo, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Lu 'an People's Hospital, Lu'an
  - Children's Hospital of Shanghai, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of Shihezi University School of Medicine, Shihezi
  - Wuhan Children's Hospital, Wuhan
- Japan (14):
  - Jinnouchi Neurosurgical Clinic, Kasuga-shi, Fukuoka
  - Ikeda Neurosurgical Clinic, Kasuga-shi, Fukuoka
  - Hikita Pediatric Clinic, Kiryu-shi, Gunma
  - Konan Medical Center, Higashinada-ku Kobe-shi, Hyōgo
  - Yamaguchi Clinic, Nishinomiya-shi, Hyōgo
  - Mito Kyodo General Hospital, Mito, Ibaraki
  - Tanaka Neurosurgery & Headache Clinic, Kagoshima, Kagoshima-ken
  - Sendai Headache and Neurology Clinic, Taihaku-ku Sendai-shi, Miyagi
  - Tennoji Dai Brain Clinic, Abeno-ku Osaka-shi, Osaka
  - Tominaga Clinic, Naniwa-ku, Osaka
  - Saitama Neuropsychiatric Institute, Chuo-ku Saitama-shi, Saitama
  - Tokyo Headache Clinic, Shibuya-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - Local lndependent Administrative Corporation Hiroshima City Hospital Organization Hiroshima City, Hiroshima
- Mexico (4):
  - Clinstile S.A. de C.V., Col. Roma Norte, Mexico City
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Clinical Reseach Institute, S.C., Tlalnepantla, State of Mexico
  - Unidad de Investigacion en Salud de Chihuahua S.C., Chihuahua City
- Poland (6):
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak, Wroclaw, Lower Silesian Voivodeship
  - NZOZ Wielospecjalistyczna Poradnia Lekarska SYNAPSIS, Lech Szczechowski, Katowice
  - Centrum Medyczne Plejady, Krakow
  - Wojewódzki Specjalistyczny Szpital Dzieciecy im. Sw. Ludwika w Krakowie, Apteka Szpitalna, Krakow
  - Clinical Research Center Sp. z.o.o. Medic-R Spolka komandytowa, Poznan
  - Euromedis Sp. z o. o., Szczecin
- Spain (6):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Centre d'Atencio Primaria Balenya, Barcelona
  - Instituto de Investigaciones del Sueno, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Sweden (3):
  - ProbarE i Lund AB, Lund, Skåne LÄN [se-12]
  - Avdelningen för kliniska Prövningar, Universitetssjukhuset Örebro, Örebro
  - ProbarE i Stockholm AB, Stockholm
- United Kingdom (3):
  - Leicester Royal Infirmary, Leicester
  - Re:Cognition Health Limited, London
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=BHV3000-311